CLINICAL TRIAL: NCT01561729
Title: Evaluation of RightBio Metrics', RightSpot pH Indicator, for Rapid Bedside Verification of Proper Nasogastric/ Orogastric Tube Placement in Emergency Department & Intensive Care Unit Patients
Brief Title: Nasogastric/Orogastric Tube Placement Verification Study Using RightSpot pH Indicator to Verify Gastric Acidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RightBio Metrics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00004691
Record Dates: First submitted 2012-01-26; First posted 2012-03-23 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Small Bowel Obstruction; Gastrointestinal Hemorrhage
Keywords: nasogastric tube; orogastric tube; RightSpot pH Indicator; suction tube; RightBio Metrics; RightLevel; RightSpot Infant; NG Tube; pH; Gastric Acidity
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): This is the only arm of the study. All patients enrolled will have a nasogastric or orogastric tube placed. All will be assessed by both the RightSpot pH Indicator and chest radiograph.
  Interventions: Device: RightSpot pH Indicator; Radiation: Chest radiograph

INTERVENTIONS:
Device: RightSpot pH Indicator — The RightSpot pH Indicator device is used to confirm proper placement of all types of gastric tubes used for gastric rest, suction, or medicating/feeding by measuring the pH of stomach aspirate. This device is intended for 1 (one) SINGLE USE. The probability of proper placement is higher when the pH is less than or equal to 4.5 and if aspirate has a typical gastric fluid appearance (grassy green, brown, colorless- with possible shreds of off-white mucus or sediment).
Radiation: Chest radiograph — Chest radiograph will be taken after tube placement to verify proper positioning of the nasogastric or orogastric tube.
  Other Names: CXR

SUMMARY:
This study will evaluate the use of RightBio Metrics' RightSpot device used to determine if there is proper placement of a nasogastric or orogastric tube.

DETAILED DESCRIPTION:
Primary objective:

To assess the level of accuracy of the RightSpot pH Indicator in determining correct placement of NG/OG tubes as compared to the gold standard of CXR in Emergency Department & ICU patients.

Hypothesis 1: In greater than 90% of the cases, RightSpot pH Indicator will be successful in confirming the placement of NG/OG tubes by demonstrating a pH of 4.5 or less in patients with CXR proven tube placement.

Hypothesis 2: The time to confirmation of NG/OG tube placement will be significantly less using the RightSpot pH Indicator than using CXR. The time will be calculated by the start time consisting of the time that the NG/OG tube was placed until the end time, which will be when the device pH Indicator testing is performed. The time to confirmation using the gold standard of a CXR will begin when the NG/OG tube is placed and end when the CXR is available on PACS (picture archiving and communication system).

Secondary objective:

To determine via subgroup analysis whether gross blood in the stomach, presence of acid-reducing medications, or trauma affects the accuracy of NG/OG placement determination by the RightSpot pH Indicator.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Patient or proxy willing to provide informed consent
* Patients who require placement of a nasogastric/orogastric tube, in the ED or ICU, as standard of care, AND a member of the study staff is available and present for NG/OG tube placement.
* It is anticipated that the patient will remain in the ED/ICU in order to obtain RightSpot pH Indicator reading and verifying CXR

Exclusion Criteria:

* Patients less than 18 years of age
* Patient or proxy unwilling or unable to provide informed consent
* Patient with known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Determination of proper placement of ng/og tube | Participants will be followed until the determination of proper placement of the ng/og tube is made. This is anticipated to be less than 3 hours.
  The pH will be assessed by visual inspection of pH paper within the device. If the pH is noted to be less than 4.5 then the placement will be considered to be within the stomach.

SECONDARY OUTCOMES:
Confounding factors for using the RightSpot pH Indicator | Participants will be followed until the determination of proper placement of the ng/og tube is made. This is anticipated to be less than 3 hours.
  A subgroup analysis will be done to determine whether gross blood in the stomach, presence of acid-reducing medications, or trauma affects the accuracy of NG/OG placement determination by the RightSpot pH Indicator.
Time to confirmation of tube placement | Participants will be followed until the determination of proper placement of the ng/og tube is made. This is anticipated to be less than 3 hours.
  The time to verification of tube placement will be measured for both chest radiograph and use of RightSpot pH Indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wilson, MD, Principal Investigator — University of South Florida Emergency Medicine Residency Program
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States